CLINICAL TRIAL: NCT07386574
Title: Testing a Contextualized and Digitalized WHO's Mental Health Action Gap Intervention Guide Substance Use Disorders Module in Primary Care Settings of Pakistan: A Feasibility Cluster Randomized Controlled Trial
Brief Title: Contextualization and Digitalization of WHO's Mental Health Action Gap Intervention Guide Substance Use Disorders Module
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Capaital University of Sceince of Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: mhGAP-IG-SUD-001; 16645 (Other Grant/Funding Number: HEC-NRPU)
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder (SUD)
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-mhGAP-IG-SUD Intervention Group (Experimental): Participants randomized to this arm will receive a total of eight bi-weekly training sessions on the use of the adapted e-mhGAP-IG-SUD-Urdu mobile application. Training will focus on improving screening, diagnosis, and management of young people with SUD and referral to specialized services where needed.
  Interventions: Other: mhGap IG SUD Module Intervention Training
- Control Group (Active Comparator): Participants randomized to this arm will continue with routine practices and standard care for SUD management as currently being delivered.
  Interventions: Other: Control

INTERVENTIONS:
Other: mhGap IG SUD Module Intervention Training — 8 bi-weekly training sessions of e-mhGAP IG SUD Module
  Arms: e-mhGAP-IG-SUD Intervention Group
Other: Control — Routine practices or standard of care
  Arms: Control Group

SUMMARY:
The aim of study is to:

1. To contextualize, adapt, customize and digitalize WHO's Mental Health Gap Action Programme Intervention Guide (e-mhGAP-IG); Substance Use Disorders Module (SUD module) V 2.0 for primary care settings (PCPs) in Pakistan.
2. To test the feasibility and acceotability of the e-mhGAP-IG (SUD module) training program in a feasibility cluster randomized controlled (cRCT) trial to enable mental health services in primary health care settings in Pakistan.

The proposed study includes contextualization, adaptation, customization, and a feasibility cRCT of e-mhGAP-IG (SUD module) V 2.0 by constituting a combination of traditional and technological approaches of eHealth (mHealth, blended learning, and telemedicine) enabling mental health services in primary care settings to be well informed and accessible. This intervention will empower 300 Primary Care Physicians (PCPs) based in Primary Care Units (PCUs) from urban settlements and Basic Health Units (BHUs) from rural settlements in three major cities, Karachi, Lahore, and Rawalpindi, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Primary and non-specialized healthcare providers working in the identified health facilities for this study across three targeted cities; willing to give informed consent for participation in this trial.

Exclusion Criteria:

* Any primary and non-specialized healthcare provider who is not permanently working in the selected health facilities, has no access to a smart mobile phone and/or internet connection; and is uncomfortable using a mobile phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility measures | From enrollement to the end of intervention at 4 weeks
  Feasibility will be determined by recruitment and retention rates of participants throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Basic Health Unit, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No